CLINICAL TRIAL: NCT03804229
Title: A Multi-center, Random, Double Blind and Placebo Control Phase III Clinical Study on the Efficacy and Safety of Butylphthalide Soft Capsule for the Treatment of Vascular Dementia
Brief Title: Efficacy and Safety of Butylphthalide Soft Capsule for the Treatment of Vascular Dementia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: CSPC-NBP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jianping Jia, Director and Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPC-NBP-2018102
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Vascular Dementia
Keywords: Vascular Dementia; cognition
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active group (Experimental): Take two pills (100 mg each) of Butylphthalide soft capsule each time, three times a day, 0.5 hours before meal, taking with lukewarm water.
  Interventions: Drug: Butylphthalide soft capsule
- control group (Placebo Comparator): Take two pills of placebo soft capsule each time, three times a day, 0.5 hours before meal, taking with lukewarm water.
  Interventions: Drug: Placebo soft capsule

INTERVENTIONS:
Drug: Butylphthalide soft capsule — 700 subjects are randomly divided into two groups by 1:1. About 350 patients in the active group take two pills(100mg each) of Butylphthalide soft capsule each time, three times a day, 0.5 hours before meal, taking with lukewarm water.
  Other Names: The effects of Butylphthalide soft capsule on VaD
  Arms: active group
Drug: Placebo soft capsule — 700 subjects are randomly divided into two groups by 1:1. About 350 patients in the active group take two pills of placebo soft capsule each time, three times a day, 0.5 hours before meal, taking with lukewarm water.
  Other Names: Placebo
  Arms: control group

SUMMARY:
Butylphthalide soft capsule has been confirmed to have beneficial effects for patients with vascular dementia (VaD) in clinical trial of phase II study. So the investigators hypothesize that Butylphthalide soft capsule may have same beneficial effects for patients with VaD in an extended samples in phase III study. In present study the investigators will recruit patients with mild to moderate VaD in a multi-center, random, double blind and placebo control methods to confirm the efficacy and safety of Butylphthalide soft capsule. The outcome measures include general cognitive function, executive function, daily living skills, and mental behavior changes of symptoms in VaD patients.

DETAILED DESCRIPTION:
Butylphthalide soft capsule is a synthetic chiral compound containing L- and D-isomers of butylphthalide. Studies in the past several decades have demonstrated that it could alleviate the learning and memory deficits induced by cerebral ischemia in rats. The phase II study enrolled 281 patients showed greater effects than placebo on ADAS-cog and CIBIC-plus. Butylphthalide soft capsule were uncommon and primarily consisted of mild gastrointestinal symptoms. In the present phase III study the investigators will re-assess the efficacy and the safety of Butylphthalide soft capsule for the treatment of mild to moderate vascular dementia in 700 subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥50 and ≤75, male or female.
* 2. The subjects must have completed primary school education or above, and be able to complete the cognitive ability test and other tests required by the program.
* 3. Meet the vascular dementia diagnosis criteria specified in the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-V).
* 4. Meet the SIVD diagnosis criteria of Erkinjuntti.
* 5. MRI supports the existence of an ischemic cerebrovascular disease; Meet the National Institute of Neurological Disorders and Stroke (NINDS-AIREN) imaging diagnosis criteria; The lesion located between supra-tentorial and subcortical areas; The maximum diameter of the infarction ≤30mm; The number of infarctions ≥3, and/or Fazekas score=2-3.
* 6. The patients need to be enrolled 3 months after the last stroke, if there is a clear history of stroke; otherwise meet other Criteria.
* 7.The subjects are suffering from mild or moderate vascular dementia, with 11≤ MMSE ≤26, and the Clinical Dementia Rating (CDR) score 1≤ CDR ≤2.
* 8. The Hamilton depression scale (HAMD) total score ≤17.
* 9. The patient agrees to participate in this study and the patient or his or her legal guardian has signed the informed consent before the study.
* 10. The subjects must have a care giver who has completed primary school education or above. The MMSE score of the care giver should be within the following range: education level of primary school > 20 points, education level above primary school > 24 points. And the care giver shall also be able to take care of the patient at least 4 days a week for more than 4 hours a day while he or she can accompany the subjects to attend each visit.

Exclusion Criteria:

* 1. Patients suffering from dementia caused by other cerebral diseases other than VaD (such as Alzheimer's disease, dementia with Lewy bodies, frontotemporal dementia, Parkinson's disease, demyelinating diseases of the central nervous system, tumors, hydrocephalus, traumas, syphilis, AIDS, Creutzfeldt-Jakob disease, etc.);
* 2. MRI indicates hippocampus or entorhinal cortex atrophy; and patients for whom VaD in combination with AD has been maximally excluded. But the following two cases can be included: ① Those aged 70 years and above with MTA score of grade 2 can be included; ② Those with grade 3 white matter injury score can be included with MTA score of grade 2.
* 3. Patients with severe neurologic impairments that hinder them from completing the required tests, such as hemiplegia of the convenient hand, various kinds of aphasia, and audio or visual disorders.
* 4. Patients who cannot swallow any orally administered drugs, or who is suffering from any disease that can affect the absorption of orally administered drugs, such as active intestinal diseases, partial or complete intestinal obstruction.
* 5. Patients suffering from severe diseases of the circulation system, the respiration system, the urinary system, the digestive system and the hemopoietic system (such as unstable angina pectoris, uncontrollable asthma and active gastric bleeding) and cancer.
* 6. Patients suffering from nutritional and metabolic diseases and endocrine system disorders, such as thyroid disease, parathyroid disease and deficiency of vitamin or other elements.
* 7. Patients suffering from severe mental diseases (such as depression and schizophrenia) and epilepsy.
* 8. Patients with alcohol or drug abuse.
* 9. Patients with a family history of dementia.
* 10. Patients who have been given any drug that can affect the cognitive function, such as cholinergic drugs, antipsychotic drugs and nootropic agents (including traditional Chinese herbal medicines and pills, such as cholinesterase inhibitors, memantine, Cenma Yizhi Capsules and Jiannaoan), for a long period of time (within 3 month before the start of this study and will continue using such drug).
* 11. Patients who have used Butylphthalide soft capsule or injection within 2 weeks before grouping.
* 12. Patients who are allergic to Butylphthalide/celery.
* 13. Patients with severe bleeding tendency or hepatic dysfunction (with transaminase higher than 3 times of the normal upper limit).
* 14. Pregnant or breast feeding women.
* 15. Patients who have participated in other interference clinical studies within 3 months before grouping.
* 16. Patients for whom MRI cranial imaging cannot be performed.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-02-07 (Estimated)

PRIMARY OUTCOMES:
Vascular Dementia Assessment Scale-cognitive Subscale(VaDAS-cog) | Change from baseline VaDAS-cog score at Week 52
  The group difference between the treatment group and the control group in the difference between the Vascular AD Assessment Scale Cognitive Subscale (VaDAS-cog) score at weeks 13, 26, 39 and 52 and the baseline score. The 6 areas of the cognitive function assessed by VaDAS-cog include the memory, the language competence, the orientation, the inferential capability, the practical ability and the comprehension. The total score is from 0 to 90 and the lower the score the milder the disease.

SECONDARY OUTCOMES:
Clinician Interview Based Impression of Severity (CIBIC-plus) | Change from baseline CIBIC-plus score at Week 52
  The group difference between the treatment group and the control group in the difference between the Clinician Interview Based Impression of Severity (CIBIC-plus) score at weeks 13, 26, 39 and 52 and the baseline score. CIBIC-plus is a kind of scale that is assessed based on the clinical changes of the patient according to the impression obtained through interviewing the patient and other insiders. The score is from 1 to 7. And 1 indicates that the recovery is optimal, 4 indicates that there is no change and 7 indicates overall worsening.
Alzheimer's Disease Co-operative Study Activities of Daily Living (ADCS-ADL) | Change from baseline ADCS-ADL score at Week 52
  The group difference in the difference between the Alzheimer's Disease Co-operative Study Activities of Daily Living (ADCS-ADL) scores at weeks 13 (±7 days), week 26 (±7 days) , week 39 (±7 days) and week 52 (±7 days) and the base line score.
Neuropsychiatric Inventory (NPI) | Change from baseline NPI score at Week 52
  It evaluates both the presence and severity of 12 neuropsychiatric features. The caregiver is asked to rate the frequency of the symptoms of that domain on a scale of 1 to 4 (1 = occasionally, less than once per week; 4 = very frequently, once or more per day or continuously) as well as their severity (1 = mild, 2 = moderate, 3 = severe). The total score for each domain is calculated by multiplying the frequency by the severity. A total score is calculated by adding all the domain scores together. Caregiver distress is rated by the caregiver on a six-point scale from 0 (no distress) to 5 (very severe or extreme distress). The total score of the caregiver's distress is obtained separately. The total NPI score is from 0 to 144 and the lower the score the milder the disease, the total caregiver distress score is from 0 to 6. The group difference between the NPI scores at weeks 13 (±7 days), week 26 (±7 days), week 39 (±7 days) and week 52 (±7 days) and the base line score.
Mini-mental State Examination (MMSE) | Change from baseline MMSE score at Week 52
  The group difference in the difference between the Mini-mental State Examination (MMSE) scores at weeks 13 (±7 days), week 26 (±7 days), week 39 (±7 days) and week 52 (±7 days) and the baseline score.
MRI | Change from baseline MRI at Week 52
  The changes before and after the treatment at the cranial MRI bilateral hippocampus, the gyrus cinguli, the posterior horn of lateral ventricle, the infarction and the frontal temporal lobe white matter volume before the treatment, and at weeks 26 (± 7days) and 52 (±7days).
Blood biomarker | Change from baseline concentration of BDNF and VEGF at Week 52
  The concentration of BDNF and VEGF measured before the treatment, and at weeks 26 (± 7days) and 52 (±7 days) respectively.
MI/Cr ratio | Change from baseline MI/Cr ratio at Week 52
  The myoinositol (MI) and the creatine (Cr) levels (obtain the MI/Cr ratio) measured before the treatment, and at weeks 26 and 52 respectively.
Acetyl choline level | Change from baseline concentration of acetyl choline at Week 52
  The concentration of acetyl choline in the blood measured before the treatment, and at weeks 26 (± 7days) and 52 (± 7days) respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, MD,PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China